CLINICAL TRIAL: NCT07189689
Title: Mental Health Mission Mood Disorder Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Oxford (Other)
Collaborators: Newcastle University (Other); University of Nottingham (Other); University of Exeter (Other); University of Southampton (Other); University of Birmingham (Other); University of Manchester (Other); University of Liverpool (Other); Avon and Wiltshire Mental Health Partnership NHS Trust (Other Government); Cambridgeshire and Peterborough NHS Foundation Trust (Other); University of Cambridge (Other); Cardiff University (Other); Cardiff and Vale University Health Board (Other Government); University of Edinburgh (Other); University of Glasgow (Other); University College, London (Other); Sheffield Health and Social Care NHS Foundation Trust (Unknown); King's College London (Other); Imperial College London (Other); Oxford Health NHS FT (Unknown); Cumbria, Northumberland, Tyne and Wear NHS FT (Unknown); South London and Maudsley NHS FT (Unknown); Nottinghamshire Healthcare NHS FT (Unknown); Devon Partnership Trust (Unknown); Hampshire and Isle of Wight Health NHS FT (Unknown); Birmingham and Solihull Mental Health NHS Trust (Unknown); Mersey Care NHS FT (Unknown); NHS Lothian (Other Government); NHS Greater Glasgow & Clyde (Unknown); Camden & Islington NHS FT (Unknown); West London NHS FT (Unknown); Central and North West London NHS FT (Unknown)
Responsible Party: Sponsor
Other Study IDs: 18955; 345799 (Other: IRAS)
Record Dates: First submitted 2025-07-31; First posted 2025-09-24 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Depression - Major Depressive Disorder; Depression Bipolar; Treatment Resistant Depression
Keywords: Observational; Cohort; Depression; UK; Mission; Bipolar; TRD; Difficult-to-treat; Treatment resistant depression; Bipolar depression; cohort study; Observational study
MeSH Terms: conditions — Bipolar Disorder; Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA, RNA, serum, plasma and peripheral blood mononuclear cells (PBMC)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current study aims to understand why some people with depression respond to treatment and others do not, using markers of clinical symptoms, both clinician reported outcome measures and patient reported outcome measures, demographic information, cognitive function, genetic sequence information (genomic), chemical measures of metabolism (metabolomic), protein makeup (proteomic) and the body's natural defence system (immune/inflammatory markers) together with collections of cells that will facilitate new research to drive improvements in diagnosis and treatment of mood disorders that may be proving difficult to treat. This will allow future clinical trials within the NHS, academia and industry to drive forward new approaches and treatments.

Participants who provide consent for re-contact for future treatment trials and other research studies have the potential to benefit from this with participation in experimental studies and clinical trials associated with improved patient outcomes. Overall, the cohort will generally support greater access to research opportunities for a wider population of people.

ELIGIBILITY:
Inclusion Criteria:

* Those aged 18 and above
* Primary clinical diagnosis of MDD or bipolar disorder based on DSM-5/ICD-11 diagnostic criteria
* Participant is willing and able to give informed consent for participation in the study
* Possesses sufficient command of the English language required to complete study requirements, as assessed by the study team

Exclusion Criteria:

* Inability to complete study activities as assessed by the study team
* Presentation requires immediate emergency treatment
* Presentation requires clinical input not available within the research clinic

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The current study aims to recruit adults aged 18 and over, currently residing in the UK with a diagnosis of major depressive disorder or bipolar disorder. The study will be advertised on social media and will allow people to self-refer to the study. We will also recruit via GP mail outs.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
PHQ-9 | Up to 36 months.
  Patient Health Questionnaire - 9-item Depression scale. Scores range between 0-27, with higher scores indicating worse depression.

OTHER OUTCOMES:
GAD-7 | Up to 36 months.
  Generalised Anxiety Disorder Questionnaire - 7 item. Scores range between 0-21, with higher scores indicating worse anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Research Facility, Warneford Hospital, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes